CLINICAL TRIAL: NCT01975818
Title: A Randomized, Parallel Group, Open-label, Multicenter Study to Investigate the Efficacy and Safety of Oral BAY85-3934 and Active Comparator (Epoetin Alfa / Beta) in the Maintenance Treatment of Subjects With Anemia Associated With Chronic Kidney Disease Who Are on Dialysis and on Treatment With an Erythropoiesis-stimulating Agent in the United States and Japan
Brief Title: Maintenance Treatment of Anemia Associated With Chronic Kidney Disease (CKD) in Hemodialysis Subjects on Epoetin Alfa / Beta Treatment Versus BAY85-3934
Acronym: DIALOGUE4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16208
Record Dates: First submitted 2013-10-18; First posted 2013-11-05 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Anemia; Renal Insufficiency, Chronic
Keywords: Anemia of CKD on dialysis
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — molidustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Molidustat (BAY 85-3934)(25mg) (Experimental): Starting dose of 25 mg of BAY85-3934 as once-daily oral tablets. Regular titrations at dose control visits. Titration occuring every 4-weeks will be based on the subject's Hb response and tolerability of the prior dose. Total treatment time is 16 weeks. Planned doses include 15, 25, 50, 75, 100,150 and 200 mg once daily.
  Interventions: Drug: Molidustat (BAY 85-3934)
- Molidustat (BAY 85-3934)(50mg) (Experimental): Starting dose of 50 mg of BAY85-3934 as once-daily oral tablets. Regular titrations at dose control visits Titration occuring every 4-weeks will be based on the subject's Hb response and tolerability of the prior dose. Total treatment time is 16 weeks. Planned doses include 15, 25, 50, 75, 100,150 and 200 mg once daily.
  Interventions: Drug: Molidustat (BAY 85-3934)
- Molidustat (BAY 85-3934) (75mg) (Experimental): Starting dose of 75 mg of BAY85-3934 as once-daily oral tablets. Regular titrations at dose control visits Titration occuring every 4-weeks will be based on the subject's Hb response and tolerability of the prior dose. Total treatment time is 16 weeks. Planned doses include 15, 25, 50, 75, 100,150 and 200 mg once daily.,
  Interventions: Drug: Molidustat (BAY 85-3934)
- Molidustat (BAY 85-3934) (150mg) (Experimental): Starting dose of 150 mg of BAY85-3934 as once-daily oral tablets. Regular titrations at dose control visits Titration occuring every 4-weeks will be based on the subject's Hb response and tolerability of the prior dose. Total treatment time is 16 weeks. Planned doses include 15, 25, 50, 75, 100, 150 and 200 mg once daily
  Interventions: Drug: Molidustat (BAY 85-3934)
- Epoetin alfa/beta (Active Comparator): Starting dose at the subject's current weekly dose. Administered IV or SC 3 times per week. Doses will be titrated at the scheduled dose control visits according to the local label. Titration will be based on the subject's Hb response and tolerability of the prior dose. Epoetin alfa may be administered in either the United States (US) or Japan; epoetin beta will only be administered in Japan.
  Interventions: Biological: Epoetin alfa/beta

INTERVENTIONS:
Drug: Molidustat (BAY 85-3934) — Oral doses of BAY85-3934 will be available in multiples of 25,50,75 and 150 mg tablets
  Arms: Molidustat (BAY 85-3934) (150mg); Molidustat (BAY 85-3934) (75mg); Molidustat (BAY 85-3934)(25mg); Molidustat (BAY 85-3934)(50mg)
Biological: Epoetin alfa/beta
  Arms: Epoetin alfa/beta

SUMMARY:
Evaluate efficacy and safety of 16 weeks of titrated dose treatment with BAY85-3934 versus epoetin alfa/beta as measured by hemoglobin (Hb) levels. Fixed starting doses of 25, 50,75 and 150 mg of BAY85-3934 titrated at the scheduled dose control visits. Titration will be based on the subject's Hb response and tolerability of the prior dose. Planned doses include 15, 25, 50, 75, 100,150 and 200 mg/day

ELIGIBILITY:
Inclusion Criteria:

* - Eligible subjects will have a diagnosis of anemia associated with CKD(chronic kidney disease).
* Women without childbearing potential
* Male or female subject ≥ 18 years of age with anemia of CKD at screening
* On dialysis, defined as regular long-term hemodialysis, with the same modality of dialysis for ≥ 3 months before randomization
* Dialysis vascular access via native arteriovenous fistula, synthetic graft, long-term catheters, or long-term tunneled catheters
* Treated with epoetin alfa (US or Japan) or epoetin beta (Japan) via intravenous (IV) or subcutaneous (SC) route, on stable dosing defined as a < 50% change from the maximum prescribed weekly dose with no change in the prescribed frequency during the last 8 weeks prior to randomization
* At least one kidney
* Mean screening Hb concentration 9.0 to 11.5 g/dL inclusive (mean of all local laboratory Hb measurements [at least 2 measurements must be taken ≥ 2 days apart] during the 4 week screening period, AND none of the measurements can be < 9.0 g/dL or > 12.0 g /dL
* Serum ferritin levels ≥ 100 μg/L OR transferrin saturation ≥ 20% at screening. Iron substitution is allowed
* Folate and vitamin B12 levels above the lower limit of normal. Supplementation is allowed
* Exclusion Criteria:
* Subjects with significant acute or chronic bleeding, such as overt gastrointestinal bleeding
* Hereditary hemoglobinopathies (including, but not limited to, sickle cell disease, beta thalassemia, and thalassemia major) which may be the primary cause of anemia
* Chronic lymphoproliferative diseases
* Any allograft (including renal allograft) in place and on immunosuppressive therapy, or a scheduled kidney transplant within the next 16 weeks (being on a waiting list does not exclude the subject)
* Chronic inflammatory disease that could impact erythropoiesis (e.g., systemic lupus erythematosis, rheumatoid arthritis, celiac disease)
* Subjects treated with immuno- or myelosuppressive therapy within 8 weeks prior to randomization: e.g., everolimus, sirolimus, rituximab, azathioprine, mycophenolate mofetil, mycophenolic acid, cyclosporine,methotrexate, and tacrolimus, chemotherapeutic agents and other anticancer agents, and systemic steroids (except inhaled steroids) for 7 days
* RBC-containing transfusion within 8 weeks before randomization
* History of cardio- (cerebro-) vascular events (e.g., unstable angina, myocardial infarction, stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within the last 6 months from the initial screening visit
* Sustained, poorly controlled arterial hypertension or hypotension at screening, defined as a mean BP ≥ 180/110 mmHg or systolic BP < 95 mmHg, respectively
* Severe rhythm or conduction disorder (e.g., HR < 50 or > 110 bpm, atrial flutter, prolonged QT >500 msec, second or third degree atrioventricular [AV]block if not treated with a pacemaker)
* New York Heart Association Class III or IV congestive heart failure
* Severe hepatic insufficiency (defined as alanine aminotransferase [ALT], aspartate aminotransferase [AST], or gamma-glutamyl transferase > 3 times the upper limit of normal [ULN], total bilirubin > 2 mg/dL, or Child-Pugh B or C) or active hepatitis in the investigator's opinion
* A scheduled surgery that may be expected to lead to significant blood loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory hemoglobin level from baseline to the average during the last 4 weeks treatment period | Baseline and weeks 14 to 17

SECONDARY OUTCOMES:
Mean of the hemoglobin (Hb) levels in the target range (10.0 to 11.0 g/dL) | From week 14 to 17
Mean of the hemoglobin levels in the target range (9.5 to 11.5 g/dL) | From week 14 to 17
Change from baseline in Hb during active treatment | Baseline and weeks 14 to 17
Number of patients with hemoglobin levels outside the target range | From week 14 to 17
Dose level in the evaluation period | Up to 16 weeks
Duration of exposure on each dose level | Up to 16 weeks
Number of subjects requiring titration of dose | Up to 16 weeks
Number of participants with serious adverse events as a measure of safety and tolerability | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- United States (24):
  - Azusa, California
  - Long Beach, California
  - Los Angeles, California
  - Lynwood, California
  - Northridge, California
  - San Dimas, California
  - Whittier, California
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - Detroit, Michigan
  - Creve Coeur, Missouri
  - Eatontown, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Fresh Meadows, New York
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Grand Prairie, Texas
  - Houston, Texas
  - Mansfield, Texas
  - San Antonio, Texas
- Japan (5):
  - Muroran, Hokkaido
  - Himeji, Hyōgo
  - Kuwana, Mie-ken
  - Kyoto
  - Nagano

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/